CLINICAL TRIAL: NCT00040144
Title: A Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Safety and Efficacy of 12 Weeks Oral Treatment With ACH126, 433 (b-L-Fd4C) in Adults With Lamivudine-resistant Chronic Hepatitis B
Brief Title: Safety and Antiviral Study of ACH126, 433 (b-L-Fd4C) in Adults With Lamivudine-resistant Chronic Hepatitis B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH443-005
Record Dates: First submitted 2002-06-21; First posted 2002-06-25 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Chronic Hepatitis B
Keywords: E-Antigen Positive; Lamivudine-resistant Chronic Hepatitis B; Achillion
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — dexelvucitabine

INTERVENTIONS:
Drug: ACH126, 433
  Other Names: b-L-Fd4C

SUMMARY:
The purpose of this study was to determine the safety and antiviral hepatitis B virus (HBV) activity of ACH126, 433 in the treatment of adults with lamivudine-resistant chronic hepatitis B.

DETAILED DESCRIPTION:
Evaluation of the safety and antiviral activity of 3 dose levels of ACH126, 433 over a 12-week treatment in the population is described.

ELIGIBILITY:
Inclusion Criteria

* Chronic HBV infection, known to be hepatitis B surface antigen (HbsAg) positive ≥ 6 months
* On lamivudine, either 100 or 150 milligrams daily for the treatment of chronic hepatitis B infection and exhibit a 2-3 log decrease in HBV deoxyribonucleic acid (DNA) levels followed by a rebound of at least 1.5 log HBV DNA or

  * Achieved an HBV DNA level of < 10,000 copies/milliliter (mL) HBV DNA on at least 2 occasions and have rebounded to > 100,000 copies/mL HBV DNA, or
  * Have a demonstrable lamivudine -resistant genotype regardless of treatment history.
* Hepatitis B e-antigen positive.
* Human immunodeficiency virus (HIV) negative.
* Serum alanine aminotransferase ≥ 1.5 and ≤ 10x times the upper limit of normal (ULN).
* Hemoglobin ≥ 10 grams/deciliter or hematocrit ≥ 30% (in the absence of blood transfusions or erythropoietin treatment in the preceding 2 weeks).
* Platelet count >75,000/cubic millimeters (in the absence of ongoing granulocyte colony-stimulating factor therapy).
* Serum creatinine < 1.1x the ULN.
* Negative radiologic screening test (ultrasound, computerized tomography scan, or magnetic resonance imaging) for hepatocellular carcinoma within 6 months prior to entry.
* Prothrombin time/international normalize ratio < 2.
* Participants of reproductive capability must utilize an approved form of birth control.
* All women of child-bearing capability must have a negative serum or urine pregnancy test (minimum sensitivity of 24 international units/liter of beta human chorionic gonadotropin) within 72 hours prior to the start of study medication.
* Participants must be able to provide written informed consent.
* Participant must be available for follow-up for a period of 20 weeks.

Exclusion Criteria

* HIV infection.
* Hepatitis C co-infection.
* Alcohol abuse.
* Pregnancy or breast-feeding.
* Inability to tolerate oral medication.
* Any clinical condition or prior therapy that, in the Investigator's opinion, would make the participant unsuitable for the study or unable to comply with the dosing requirements.
* Use of any investigational drug.
* Participants with decompensated liver disease.
* Use of any concomitant herbal treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Start 2002-07; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (11):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, Pasadena, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Fairfax, Virginia
  - Clinical Trial Site, Seattle, Washington
- Canada (3):
  - Clinical Trial Site, Vancouver, British Columbia
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Montreal, Quebec
- Clinical Trial Site, Hong Kong, China